CLINICAL TRIAL: NCT05642455
Title: A Phase 1/2 Open Label, Basket Study to Assess the Safety, Tolerability and Anti-Tumor Activity of Afamitresgene Autoleucel in Pediatric Subjects With MAGE-A4 Positive Tumors
Brief Title: SPEARHEAD-3 Pediatric Study
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: USWM CT, LLC (Industry)
Responsible Party: Sponsor
Organization: USWM, LLC (dba US WorldMeds) (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADP-0044-004
Record Dates: First submitted 2022-11-07; First posted 2022-12-08 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Synovial Sarcoma; Malignant Peripheral Nerve Sheath Tumor (MPNST); Neuroblastoma (NBL); Osteosarcoma
MeSH Terms: conditions — Sarcoma, Synovial; Neurofibrosarcoma; Neuroblastoma; Osteosarcoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Afamitresgene autoleucel (Experimental)
  Interventions: Genetic: Afamitresgene autoleucel

INTERVENTIONS:
Genetic: Afamitresgene autoleucel — Single infusion of afamitresgene autoleucel Dose: For subjects ≥10 kg to <40 kg: starting dose of 0.025 - 0.200 x 10'9 transduced cells/kg. For subjects ≥40 kg 1.0x109 to 10x109 transduced by a single intravenous infusion

SUMMARY:
This is a pediatric basket study to investigate the safety and efficacy of afamitresgene autoleucel in HLA-A*02 eligible and MAGE-A4 positive subjects aged 2-17 years of age with advanced cancers.

ELIGIBILITY:
Inclusion Criteria:

* Subject has histologically confirmed diagnosis of any one of the following cancers: (A) Synovial Sarcoma (SS), (B) MPNST, (C) Neuroblastoma, or (D) Osteosarcoma (OS).
* Age:

(A) Synovial Sarcoma: 2 to 17 years (B) MPNST, Neuroblastoma and Osteosarcoma: 2 to 21 years

* Body weight ≥ 10 kg
* Must have previously received a systemic chemotherapy
* Measurable disease prior to lymphodepletion according to RECIST v1.1 (or INCR, 2017 Neuroblastoma only).
* HLA-A*02 positive
* Tumor shows MAGE-A4 expression confirmed by central laboratory.
* Performance Status:

(A) Subjects ≥16: Eastern Cooperative Oncology Group (ECOG) 0 or 1 (B) Subjects 2 to 16: Lansky score ≥ 80

• Subject has anticipated life expectancy of greater than 3 months in the opinion of the investigator.

Exclusion Criteria:

* Positive for HLA-A*02:05 in either allele; or any A*02 having same protein sequence as HLA-A*02:05
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to fludarabine, cyclophosphamide.
* History of autoimmune or immune mediated disease
* Known central nervous system (CNS) metastases.
* Other prior malignancy that is not considered by the Investigator to be in complete remission
* Clinically significant cardiovascular disease
* Active infection with human immunodeficiency virus, hepatitis B virus, hepatitis C virus, or human T cell leukemia virus
* Pregnant or breastfeeding
* Experiencing ongoing rapid disease progression that in the opinion of the Investigator significantly increases the subjects risk associated with treatment.

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2038-07-30 (Estimated)

PRIMARY OUTCOMES:
Incidence, duration, and severity of Treatment Emergent Adverse Events as assessed by Investigator Evaluation. | 3.5 years
  Determination of incidence, severity and duration of adverse events
  * Incidence of dose limiting toxicities DLTs
  * AEs including serious adverse events (SAEs)
  * Incidence, severity, and duration of the AEs of special interest
  * Replication competent lentivirus (RCL)
  * T-cell clonality and insertional oncogenesis (IO)

SECONDARY OUTCOMES:
Efficacy: Objective response rate (ORR) assessed by investigator per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 (or by International Neuroblastoma Response Criteria [INRC] 2017 in Neuroblastoma subjects) | 3.5 years
  ORR is defined as incidence of complete responses or partial responses as assessed by RECIST v1.1 or INRC, 2017
Time to response (TTR) | 3.5 years
  For patients who are observed to respond to afamitresgene autoleucel in the time from date of infusion to achieve a partial response or complete response (TTR) is assessed
Duration of Response (DoR) | 3.5 years
  For patients who are observed to respond to afamitresgene autoleucel the DoR is the date of initial response (including confirmation) from date of infusion up until disease progression
Best overall response (BOR) | 3.5 years
  BOR is assessed by the investigator per RECIST V1.1 or INCR, 2017 (for Neuroblastoma subjects)
Progression Free Survival (PFS) | 3.5 years
  PFS is assessed by the investigator from date of infusion of ADP-A2M4 up until the date of disease progression per RECIST v1.1 or death.
Overall Survival (OS) | 15 years
  OS is assessed from date of infusion of ADP-A2M4 up until the date of patient death.
Characterize the in vivo cellular pharmacokinetics (PK) profile of afamitresgene autoleucel by evaluation of PBMC samples for peak persistence. | 3.5 years
  Obtain PBMC samples for the evaluation of peak persistence of afamitresgene autoleucel.
Development and validation of an invitro diagnostic (IVD) assay for the screening of tumor antigen expression for regulatory approval. | 3.5 years
  Retention of additional tumor tissue during Pre-Screening to enable development and validation of a MAGE-A4 antigen expression companion diagnostic (CDx) assay.

CONTACTS AND LOCATIONS:
Overall Officials: Fiorella Iglesias Cardenas, MD, Principal Investigator — Memorial Sloan Kettering Kids
Locations (10):
- United States (10):
  - Stanford University, Palo Alto, California
  - National Institutes of Health, Bethesda, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Memorial Sloan Kettering Kids, New York, New York
  - Duke University School of Medicine, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philedephia, Philadelphia, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington
  - University of Wisconsin Cancer Center, Madison, Wisconsin